CLINICAL TRIAL: NCT01598376
Title: A Prospective Double-blind Interventional Study of Tissue Reaction to Polyglycolic Acid Sutures in Human Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Principal Investigator, Ben Parkin, Consultant Ophthalmologist, The Royal Bournemouth Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RBH Suture Study
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Lower Eyelid Entropion
Keywords: entropion; suture; granuloma; tissue reaction
MeSH Terms: conditions — Entropion; Granuloma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5/0 gauge vicryl suture (Active Comparator): Patients randomly assigned to 5/0 gauge test everting suture
  Interventions: Procedure: 5/0 vicryl test suture
- 7/0 gauge vicryl suture (Active Comparator): Patients randomly assigned to 7/0 gauge test everting suture
  Interventions: Procedure: 7/0 vicryl suture

INTERVENTIONS:
Procedure: 7/0 vicryl suture — 7/0 vicryl test suture placed as one of 3 everting sutures
  Arms: 7/0 gauge vicryl suture
Procedure: 5/0 vicryl test suture — 5/0 vicryl test suture placed as one of 3 everting sutures
  Arms: 5/0 gauge vicryl suture

SUMMARY:
Objective

To investigate the tissue reaction produced by implanted polyglactin suture material in normal human skin and to determine the effect of suture gauge on this response.

Design

A prospective, double blind, randomized clinical trial using a novel ethical study design. Both the patient and clinician analyzing the histology were blinded to the suture gauge used.

Participants

A total of 42 consecutive patients presenting to an oculoplastic clinic with involutional entropion and horizontal eyelid laxity, who provided written consent to participate, were enrolled in the study.

Intervention

Patients were randomly allocated to 5/0 or 7/0 Vicryl™ test suture groups. Patient symptoms were alleviated during the wait for definitive surgery by the placement of temporary eyelid everting sutures including a test suture. After 28 days, entropion correction was achieved by a Quickert procedure which includes excision of an eyelid wedge. Histological analysis was carried out, blind to the suture gauge used, on the excised eyelid containing the test suture.

Main outcome measure

Defined histological parameters of suture-related granulomas were measured at multiple levels. Data included granuloma outer diameter, central cellular diameter, giant cell number and area of fibrous coat (calculated from the coat diameter and thickness at multiple levels) and a statistical comparison made between the 5/0 and 7/0 suture gauge groups.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients
* Involutional lower eyelid entropion
* Horizontal eyelid laxity associated
* Informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Previous eyelid surgery
* Poorly controlled diabetes
* Oral steroid use
* Addisons disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Suture associated granuloma outer diameter | 28 days
  Histological measurement of suture associated granuloma outer diameter on excised eyelid specimens, average of 6 sections examined
Suture associated granuloma central cellular element diameter | 28 days
  Histological measurement of suture associated granuloma central cellular element diameter on excised eyelid specimens, average of 6 sections examined
Suture associated granuloma fibrous coat area | 28 days
  Histological measurement of suture associated granuloma fibrous coat area on excised eyelid specimens, average of 6 sections examined
Suture associated granuloma giant cell number | 28 days
  Count of giant cells on average of 6 histological sections from excised eyelid specimens

CONTACTS AND LOCATIONS:
Overall Officials: Ben Parkin, MD, Principal Investigator — Royal Bournemouth Hospital
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom